CLINICAL TRIAL: NCT04035447
Title: Improving Symptom Management for Survivors of Young Adult Cancer
Brief Title: Symptom Management for YA Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00103249; 1K08CA245107-01 (NIH)
Record Dates: First submitted 2019-07-24; First posted 2019-07-29 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Young Adult; Pain; Psychological Distress; Fatigue; Breast Cancer; Melanoma; Hematologic Cancer; Germ Cell Tumor; Endocrine Cancer
Keywords: Cancer; Young Adult; Behavioral Symptom Management
MeSH Terms: conditions — Neoplasms; Pain; Fatigue; Breast Neoplasms; Melanoma; Hematologic Neoplasms; Neoplasms, Germ Cell and Embryonal; Endocrine Gland Neoplasms

STUDY DESIGN:
Intervention Model Description: A two-arm, pilot RCT employing a wait-list control arm will be used. Six cohorts of YA survivors (n=10/cohort) are randomized within their cohort with equal allocation to the intervention or control arms. Randomization was stratified by gender.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Symptom Management for Young Adult Cancer Survivors (Experimental): The intervention provides systematic training in cognitive and behavioral coping skills (e.g., activity-rest cycling, cognitive defusion, relaxation training) delivered over the course of 8 sessions (12 therapy hours). By employing these strategies, participants learn to adjust their behaviors and emotions as well as interact differently with their thoughts in the service of better managing symptoms.
  Interventions: Behavioral: Behavioral Symptom Management for Young Adult Cancer Survivors
- Waitlist Control (Active Comparator): Waitlist control participants will receive the intervention and receive systematic training in cognitive and behavioral coping skills approximately 6 months into their participation in the study.
  Interventions: Behavioral: Behavioral Symptom Management for Young Adult Cancer Survivors

INTERVENTIONS:
Behavioral: Behavioral Symptom Management for Young Adult Cancer Survivors — The intervention includes group sessions held over Zoom along with an integrated mobile application to provide participants with instruction in cognitive and behavioral strategies for managing symptoms (i.e., pain, fatigue, distress). The developed intervention includes 8 face-to-face group sessions (12 therapy hours). Sessions are delivered using a faded contact approach (i.e., sessions 1-6: weekly, sessions 7-8: biweekly). Participants receive secure access to a study-specific mobile application that includes: 1) audio and video files and brief text-based educational content reviewing strategies discussed during the groups; 2) the ability to self-monitor symptom severity; 3) the ability to connect with group members via a social networking platform; and 4) activity tracking synchronization.

SUMMARY:
Symptom interference is common for survivors of young adult cancer (aged 18-39 at diagnosis) and impacts their abilities to achieve normative life goals (e.g., education, careers, independence, romantic/social relationships) as well as adhere to recommended follow-up care. Assistance with symptom management has been rated by young adult survivors as an important and unmet healthcare need; however, skill-based symptom management interventions have typically been tested among older cancer survivors and have not targeted the unique developmental needs of those diagnosed as young adults. The proposed research advances the health and wellbeing of young adult cancer survivors by creating a developmentally appropriate hybrid in-person/mHealth behavioral symptom management intervention which addresses variables (i.e., symptoms and symptom interference) consistently linked to significant social, economic, and health burden.

DETAILED DESCRIPTION:
More than 60,000 young adults (YAs) aged 18-39 are diagnosed with cancer in the US each year. Advances in treatment have yielded five year survival rates >70% suggesting that the majority of YAs will become long-term cancer survivors. Symptom (e.g., pain, fatigue, distress) interference is common for YA cancer survivors and impacts their abilities to achieve normative life goals (e.g., returning to work/school, achieving autonomy, pursuing social/romantic relationships) and adhere to recommended follow-up care. Symptom management has been identified as a significant issue in the transition to survivorship for YAs by the Institute of Medicine and National Cancer Institute, and assistance with symptom management is rated as an important and unmet need by YA survivors. Yet, behavioral symptom management interventions have not targeted the needs of those diagnosed as YAs. The proposed study aims to develop and test the feasibility and acceptability of a novel behavioral symptom management intervention designed for survivors of YA cancer (cancer types: hematologic, breast, or gastrointestinal cancers, melanoma, or germ cell tumors). The hybrid intervention will include inperson, group sessions and an integrated mobile application. The intervention will provide peer support while also teaching skills to improve symptoms, symptom interference, and self-efficacy for symptom management. The mobile application will assist with symptom monitoring, home skills practice, and connecting with group members. The preliminary version of the intervention will be guided by the research team's prior work developing and testing symptom management interventions for cancer survivors, national guidelines for YA oncology, consultation with an expert advisory board, and input from patient (n=20) and provider N=10) stakeholders. The intervention will be further refined following review by patient user testers (n=10). Next, feasibility, acceptability, and distributions of change over time as well as relationships between outcome variables will be examined through a pilot randomized clinical trial of the developed intervention. Participants (N=60) will be randomized to intervention or wait-list control arms. Primary study outcomes are symptom (pain, fatigue, distress) severity and symptom interference. Self-efficacy and support will also be examined as mediators of change in outcome variables. The proposed study has the potential to make several significant contributions by targeting an underserved group of cancer survivors, addressing a critical gap in care, and addressing variables consistently linked to social, economic, and health burden for YAs. It will also provide important information about approaches to identify, recruit, and retain YA cancer survivors in research and provide pilot data for a larger trial.

ELIGIBILITY:
Young Adult Cancer Survivors Participating in Intervention Development Interviews

Eligibility Criteria

* Diagnosed with hematologic, breast, gastrointestinal, or endocrine cancers, melanoma, or germ cell tumors
* Diagnosed with cancer as a young adult
* Under the care of a medical provider at the Duke Cancer Institute
* Completed curative treatment involving multimodal therapy within the last five years
* Able to speak and read English
* Able to give informed consent

Exclusion Criteria

* Nonambulatory
* Major mental illness, i.e., schizophrenia
* Untreated or uncontrolled mental illness, i.e., bipolar
* Residence greater than 100 miles from the research site

Medical Providers Participating in Intervention Development Interviews Eligibility criteria

o Provide care to young adult cancer survivors at the Duke Cancer Institute

Young Adult Cancer Survivor User Testers

Eligibility Criteria

* Diagnosed with hematologic, breast, gastrointestinal cancers, or endocrine cancers, melanoma, or germ cell tumors
* Diagnosed with cancer as a young adult
* Under the care of a medical provider at the Duke Cancer Institute
* Completed curative treatment involving multimodal therapy within the last five years
* Able to speak and read English
* Able to give informed consent

Exclusion Criteria

* Nonambulatory
* Major mental illness, i.e., schizophrenia
* Untreated or uncontrolled mental illness, i.e., bipolar
* Residence great than 100 miles from the research site

RCT Participants

Eligibility Criteria:

* diagnosed with cancer as a YA (aged 18-39)
* diagnosis of hematologic, breast, endocrine or gastrointestinal cancer, melanoma, or germ cell tumor
* receiving care at the Duke Cancer Institute
* completed curative treatment involving multimodal therapy within the last 2 years
* able to speak/read English; and able to give informed consent.

Exclusion Criteria:

* non-ambulatory
* major mental illness (i.e., schizophrenia)
* untreated or uncontrolled mental illness (i.e., bipolar disorder)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caroline S Dorfman, Principal Investigator — Duke University
Locations (1):
- Duke Cancer Institute, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dorfman CS, Shelby RA, Stalls JM, Thomas SM, Arrato NA, Herold B, Somers TJ, Keefe FJ, Winger JG, Vilardaga JP, Oeffinger K. Improving symptom management for survivors of young adult cancer: rationale and study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2024 Jun 8;10(1):87. doi: 10.1186/s40814-024-01510-7. PMID 38851732
- [Derived] Dorfman CS, Shelby RA, Stalls JM, Somers TJ, Keefe FJ, Vilardaga JP, Winger JG, Mitchell K, Ehren C, Oeffinger KC. Improving Symptom Management for Survivors of Young Adult Cancer: Development of a Novel Intervention. J Adolesc Young Adult Oncol. 2023 Aug;12(4):472-487. doi: 10.1089/jayao.2022.0100. Epub 2022 Sep 30. PMID 36178972

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a comprehensive cancer center.
Pre-assignment Details: Of 65 enrolled patients, 4 patients were excluded prior to randomization: two lost to follow up, one subject withdrawal, and one PI withdrawal due to disease progression.
Units Other Than Participants: Cohorts
Period: Treatment Period
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Started | 31; 3 Cohorts | 30; 3 Cohorts
Completed | 25; 3 Cohorts | 23; 3 Cohorts
Not Completed | 6; 0 Cohorts | 7; 0 Cohorts
Not completed — Lost to Follow-up | 6 | 5
Not completed — Physician Decision | 0 | 2
Period: Waitlist Cross-over
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Started | 27; 3 Cohorts | 0; 0 Cohorts
Completed | 27; 3 Cohorts | 0; 0 Cohorts
Not Completed | 0; 0 Cohorts | 0; 0 Cohorts

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 33 [28 to 36] | 34 [30.5 to 36] | 34 [29 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 29 | 27 | 56
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 24 | 20 | 44
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 30 | 61

OUTCOME MEASURES:

1. Primary Outcome: Intervention Satisfaction: Satisfaction With Therapy and Therapist Scale-Revised (STTS-R)
Description: Intervention satisfaction will be assessed using the Satisfaction witth Therapy and Therapist Scale-Revised, a 13-item measure with the first 12-items on a five-point scale ranging from 1 "strongly disagree" to 5 "strongly agree." The 13th item (Global Improvement) asks, "How much did the intervention help with your symptoms?" with 5 answer choices ranging from "made things a lot better" (1) to "made things a lot worse" (5). Each of the subscales (Satisfaction With Therapy and Satisfaction With Therapist) range from 6 to 30, with higher scores indicating greater overall satisfaction. A total score is calculated as the sum of the first twelve items, with possible scores from 12 to 60, with higher scores indicating greater overall satisfaction.
Time Frame: Following completion of the intervention, up to 12 months
Population: Participants who completed at least one intervention session.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Number analyzed (Participants) | 28 | 24
scores on a scale
  Satisfaction With Therapy (ST) | 26.71 (3.52) | 27.33 (3.14)
  Satisfaction With Therapist (SWT) | 28.86 (1.86) | 27.75 (3.27)
  Global Improvement (Item 13) | 1.75 (0.52) | 1.58 (0.65)
Statistical Analysis 1: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; Satisfaction with Therapy (ST); Test type: Superiority; p = 0.519, t-test, 2 sided
Statistical Analysis 2: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; Satisfaction with Therapist (SWT); Test type: Superiority; p = 0.150, t-test, 2 sided
Statistical Analysis 3: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; Global Improvement (Item 13); Test type: Superiority; p = 0.309, t-test, 2 sided

2. Primary Outcome: Number of Participants Who Completed Open-Ended Questions About the Program
Description: Intervention will be evaluated using 3 open-ended questions, including the following: "1) What was the most helpful part of the program?," "2) What was the least helpful part of the program?", and "3) What suggestions do you have for us to help improve the program?"
Time Frame: Following completion of the intervention, up to 12 months
Population: Participants who completed at least one intervention session.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Number analyzed (Participants) | 28 | 24
Participants | 28 | 24

3. Primary Outcome: Percentage of Sessions Attended by Each Participant
Description: Treatment feasibility will be assessed by measuring the session attendance rate for each participant.
Time Frame: Following completion of the intervention, up to 12 months
Population: Any participant who had at least one intervention session was included for analysis.
Measure: Mean (Standard Deviation); unit: percentage of sessions
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Number analyzed (Participants) | 28 | 27
percentage of sessions | 91.96 (23.87) | 94.27 (18.42)
Statistical Analysis 1: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; Test type: Superiority; p = 0.696, t-test, 2 sided

4. Primary Outcome: Treatment Acceptability Questionnaire
Description: The Treatment Acceptability Questionnaire is a six-item scale assessing participants' views of an intervention as acceptable, ethical, and effective. Items are rated on a 7-point Likert scale (e.g., 1 "very unacceptable" to 7 "very acceptable") and averaged.
Time Frame: Following completion of the intervention, up to 12 months
Population: One participant in the waitlist control condition was excluded from analysis due to an incomplete response to the measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Number analyzed (Participants) | 28 | 23
score on a scale | 6.54 (0.41) | 6.36 (0.83)
Statistical Analysis 1: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; Test type: Superiority; p = 0.350, t-test, 2 sided

5. Primary Outcome: Use of Intervention Strategies
Description: Participants' use of intervention strategies will be assessed using a measure developed specific to components of the proposed intervention. Participants will be asked about how frequently treatment strategies discussed in session have been used outside of session since the previous session or last assessment depending on the timing of the questionnaire. A scale ranging from 0 "not at all" to 5 "every day" will be used.
Time Frame: Following completion of the intervention, up to 12 months
Population: Any participant who had at least one intervention session was included for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Number analyzed (Participants) | 28 | 27
score on a scale | 2.35 (0.83) | 2.67 (1.24)
Statistical Analysis 1: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; Outcomes were compared at post-intervention visit: 3-month (A2) for intervention participants, 9-month (A4) for waitlist control participants; Test type: Superiority; p = 0.274, Fisher Exact

6. Primary Outcome: Self-reported Use of the Mobile Application
Description: Participants' use of the mobile application will be assessed using a measure developed specific to components of the proposed mobile application. Participants will be asked about how frequently they have used components of the mobile application outside of session since the previous session or last assessment depending on the timing of the questionnaire. A scale ranging from 0 "not at all" to 5 "2 or more times a day" will be used.
Time Frame: Following completion of the intervention, up to 12 months
Population: Any participant who had at least one intervention session was included for analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control
Number analyzed (Participants) | 28 | 27
score on a scale | 0.79 (0.9) | 0.96 (1.37)
Statistical Analysis 1: Comparison: Behavioral Symptom Management for Young Adult Cancer Survivors vs Waitlist Control; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.600, Fisher Exact

7. Secondary Outcome: Change in Depressive Symptoms: PROMIS Depression Short Form
Description: Depressive Symptoms will be assessed using the Patient Reported Outcomes Measurement Information System Depression Short Form-8a, an 8-item measure assessing symptoms of depression in the last week. Participants are asked to respond to items (e.g., "I felt sad," "I felt helpless") using a five-point scale ranging from 1 "never" to 5 "always." Items are summed and converted to standardized t-scores with a mean of 50 and standard deviation of 10. Higher T-scores indicate higher levels of depression. T-scores of 55 to 60 indicate mild levels of depression, 60 to 70 indicates moderate levels of depression, and greater than 70 indicate severe levels of depression.
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment, pre-intervention (baseline for Intervention, 6 months for Waitlist Control) and post-intervention (3 months for Intervention, 9 months for Waitlist Control) reported
Population: Respondents were included if they provided a complete response to the measure. All participants received the intervention.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- Pre-Intervention: Pre-intervention responses for participants assigned to all conditions. This group includes responses at baseline (A1) for participants assigned to Behavioral Symptom Management and 6 months (A3) for participants assigned to waitlist control.
- Post-Intervention: Responses immediately following intervention delivery for participants assigned to all conditions. This group includes responses at 3 months (A2) for participants assigned to Behavioral Symptom Management and 9 months (A4) for participants assigned to waitlist control.
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 60 | 55
T-score | 50.3 (10.2) | 48.7 (9.6)
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority; p = 0.1848, Wilcoxon (Mann-Whitney); Effect size (Hedges' g) of 0.18; Mean Difference (Net) = 1.5, Standard Deviation 8.4

8. Secondary Outcome: Change in Anxiety: PROMIS Anxiety Short Form
Description: Symptoms of Anxiety will be assessed using the Patient Reported Outcomes Measurement Information System Anxiety Short Form-8a, an 8-item measure assessing symptoms of anxiety in the last week. Participants are asked to respond to items (e.g., "I felt nervous," "I felt tense") using a five-point scale ranging from 1 "never" to 5 "always". Total scores are then converted to T-scores. Items are summed and converted to standardized t-scores with a mean of 50 and standard deviation of 10. Higher T-scores indicate higher levels of anxiety. T-scores of 55 to 60 indicate mild levels of anxiety, 60 to 70 indicates moderate levels of anxiety, and greater than 70 indicate severe levels of anxiety.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 60 | 55
T-score | 53.1 (12) | 52.6 (12)
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority; p = 0.6153, Wilcoxon (Mann-Whitney); Effect size (Hedges' g) of 0.07; Mean Difference (Net) = 0.6, Standard Deviation 8.4

9. Secondary Outcome: Change in Symptom Interference: Illness Intrusiveness Rating Scale
Description: Symptom interference will be assessed using the Illness Intrusiveness Rating Scale (IIRS). The IIRS assesses the extent to which an illness and/ or its treatments interfere with 13 quality of life domains (e.g., health, diet, work, sex life, active recreation). Items are rated on a 7-point scale from 1 "not very much" to 7 "very much." The total score ranges from 7 to 91, where a higher score indicates greater interference.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 57 | 48
score on a scale | 36.4 (20) | 32.8 (17.4)
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority; p = 0.0563, Wilcoxon (Mann-Whitney); Effect size (Hedges' g) of 0.28; Mean Difference (Net) = 4.6, Standard Deviation 16.1

10. Secondary Outcome: Change in Pain: Brief Pain Inventory
Description: The Brief Pain Inventory is a 9-item, self-report measure assessing pain severity and interference from pain across important life domains (e.g., general activity, work, relations with others). Participants rate their pain on a scale from 0 "no pain" to 10 "pain as bad as you can imagine." Pain severity is calculated as the average of four items assessing participants' worst, least, current, and average (in the last week) pain on a scale from 0 "no pain" to 10 "worst pain." Pain interference is computed as the average of seven items, which ask about the interference of pain across different life domains (e.g., general activity, mood, relations with other people).
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment; pre-intervention (baseline for Intervention, 6 months for Waitlist Control) and post-intervention (3 months for Intervention, 9 months for Waitlist Control) reported
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 60 | 52
score on a scale
  Pain Severity | 2.1 (2) | 1.7 (1.9)
  Pain Interference: number analyzed (Participants) | 58 | 48
  Pain Interference | 2.2 (2.3) | 1.9 (2.3)
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority; p = 0.0265, Wilcoxon (Mann-Whitney); Effect size (Hedges' g) of 0.31; Mean Difference (Net) = 0.6, Standard Deviation 1.8
Statistical Analysis 2: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority; p = 0.2084, Wilcoxon (Mann-Whitney); Effect size (Hedges' g) of 0.18; Mean Difference (Net) = 0.5, Standard Deviation 2.6

11. Secondary Outcome: Change in Fatigue: PROMIS Fatigue Short Form
Description: Fatigue will be assessed using the Patient Reported Outcomes Measurement Information System Fatigue Scale, a 6-item self-report measure of fatigue. Participants are asked to think about the last week when responding to each item (e.g., "In the past 7 days, how run-down did you feel, on average?"). Items are summed and converted to standardized t-scores with a mean of 50 and standard deviation of 10. A higher score indicates greater fatigue. T-scores of 55 to 60 indicate mild levels of fatigue, 60 to 70 indicates moderate levels of fatigue, and greater than 70 indicate severe levels of fatigue.
Time Frame: as for outcome 7
Population: All participants received the intervention.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Pre-Intervention | Post-Intervention
Number analyzed (Participants) | 60 | 55
T-score | 54 (10.8) | 55.4 (9.3)
Statistical Analysis 1: Comparison: Pre-Intervention vs Post-Intervention; Test type: Superiority; p = 0.3512, Wilcoxon (Mann-Whitney); Effect size (Hedges' g) of -0.13; Mean Difference (Net) = -1.2, Standard Deviation 9.4

12. Other Pre Specified Outcome: Change in Activity: International Physical Activity Questionnaire
Description: The International Physical Activity Questionnaire is a seven-item questionnaire that assesses the amount of time participants have spent doing physical activity (e.g., moderate physical activities, vigorous physical activities, walking) in the last seven
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

13. Other Pre Specified Outcome: Change in Activity: Stanford Leisure-Time Activity Categorical Item (LCAT)
Description: The Stanford LCAT is a categorical item that assesses the type of physical activities participants do.
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

14. Other Pre Specified Outcome: Change in Spritual Well-Being: Functional Assessment of Chronic Illness Therapy (FACIT)
Description: The FACIT assesses the spiritual wellbeing of participants with 12-item questionnaire on a scale from 0 = "not at all" to 4 = "very much."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

15. Other Pre Specified Outcome: Changes in Cancer Experience: Acceptance and Action Questionnaires for Cancer (AAQ)
Description: The AAQ is a 7-item questionnaire to track psychological flexibility related to coping with cancer and cancer treatment. The scale ranges from 1 = "never true" to 7 "always true." Item is scored by adding all of the responses together.
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

16. Other Pre Specified Outcome: Changes in Living in Alignment With Values: The Valuing Questionnaire (VQ)
Description: The VQ is a 10-item self-report questionnaire with a scale 0 = "not true at all" to 6 "completely true."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

17. Other Pre Specified Outcome: Group Therapy Experiences Scale
Description: The 17-item Group Therapy Experiences Scale will be used to assess the level of cohesion among group members (e.g., development of positive relationships, comfort level with other group members). Items 1-16 are rated on a 5-point scale with 1 = "strongly agree" to 5 = "strongly disagree." Item 17 is an open-ended question, "was there something in the group today that helped or hindered you?"relationships, comfort level with other group members). Items are rated on a 4-point scale with 1= "strongly disagree" to 4= "strongly agree."
Time Frame: Following completion of the intervention, up to 12 months
Reporting Status: Not Posted, anticipated posting 2025-08

18. Other Pre Specified Outcome: Change in Social Isolation: PROMIS Social Isolation Scale
Description: The PROMIS Social Isolation Scale is a 6-item measure is used to assess social isolation. Participants are asked to rate each item (e.g., "I felt left out," "I feel that people avoid talking to me") on a scale from 1= "never" to 5= "always."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

19. Other Pre Specified Outcome: Change in Self-Efficacy: The Self-Efficacy for Managing Chronic Disease Scale
Description: The Self-Efficacy for Managing Chronic Disease Scale is a 6-item scale. Participants rate their confidence in keeping pain, fatigue, emotional distress, and other symptoms from interfering with things they want to do on a scale from 1 "not at all confident" to 10 "totally confident."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

20. Other Pre Specified Outcome: Change in Self-Efficacy: PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 4a
Description: The PROMIS Self-Efficacy for Managing Chronic Conditions - Managing Symptoms - Short Form 4a is a 4-item scale. Participants rate their confidence in managing their symptoms during daily activities, with relationships with friends and family, in a public place, and working with their doctor to manage these symptoms on a scale from 1 = "I am not at all confident" to 5 "I am very confident."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

21. Other Pre Specified Outcome: Change in Emotional Support: PROMIS Emotional Support-Short Form
Description: The PROMIS Emotional Support Short Form is a 6-item measure used to assess emotional support. Participants are asked to rate each item ("I have someone who will listen to me when I need to talk," "I have someone to talk with when I have a bad day") on a scale from 1= "never" to 5= "always."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

22. Other Pre Specified Outcome: Change in Instrumental Support: PROMIS Instrumental Support-Short Form
Description: The PROMIS Instrumental Support Short Form is a 6-item measure used to assess instrumental support. Participants are asked to rate each item (e.g., "Do you have someone to take you to the doctor if you needed it?," "Do you have someone to prepare your meals if you are unable to do it yourself?") on a scale from 1= "never" to 5= "always."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

23. Other Pre Specified Outcome: Change in Informational Support: PROMIS Informational Support-Short Form
Description: The PROMIS Informational Support Short Form is a 6-item measure used to assess informational support. Participants are asked to rate each item (e.g., "I have someone to turn to for suggestions about how to deal with a problem," "I have someone to give me information if I need it") on a scale from 1= "never" to 5= "always."
Time Frame: Baseline and again 3, 6, 9, and 12 months following the baseline assessment
Reporting Status: Not Posted, anticipated posting 2025-08

ADVERSE EVENTS:
Time Frame: From enrollment until end of follow-up, up to 12 months
Groups:
- Waitlist Control - Intervention; Waitlist Control - No Intervention: Waitlist control participants will receive the intervention and receive systematic training in cognitive and behavioral coping skills approximately 6 months into their participation in the study.
Arm/Group | Behavioral Symptom Management for Young Adult Cancer Survivors | Waitlist Control - Intervention | Waitlist Control - No Intervention
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/27 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/27 | 0/3
Other Adverse Events (participants affected / at risk) | 0/31 | 0/27 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-30): https://cdn.clinicaltrials.gov/large-docs/47/NCT04035447/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT04035447/ICF_000.pdf